CLINICAL TRIAL: NCT06224881
Title: Treating Vitamin C Deficiency in Septic Shock: Would it Help?
Brief Title: Vitamin C Deficiency in Septic Shock
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Farouk, Lecturer of critical care, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MS-362-2019
Record Dates: First submitted 2023-12-28; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin C group (Active Comparator): Ascorbic acid (Vitamin C) was given parenterally (2 gm every 8hrs) for 4 days.
  Interventions: Drug: Ascorbic acid
- Control group (Placebo Comparator): No vit C given
  Interventions: Drug: Ascorbic acid

INTERVENTIONS:
Drug: Ascorbic acid — 2 gm every 8hrs for 4 days

SUMMARY:
Objectives: investigators aim to study the effect of addition of vitamin C as a part of treatment in septic shock patients on: Hemodynamics, Inflammation status and ICU outcome.

Subjects and methods: A prospective interventional randomized cohort study, was conducted on 150 consecutive patients who were admitted to the ICU with septic shock based on SIRS, SOFA and APACHE II. Treatment group (n=75) had given ascorbic acid (Vitamin C) parenterally 6gm daily and control group (n=75). Measuring the level of Vitamin C in all study population (normal range 50-70 μM/L) before and after period of 4 days.

DETAILED DESCRIPTION:
AIM OF THE WORK investigators aim to study the effect of addition of vitamin C in septic shock patients on:

* Mean arterial pressure
* C-reactive protein as an inflammatory marker
* Vasopressors ( norepinephrine) dose and duration.
* ICU outcome ( ICU stay, 7 and 28 days mortality)

SUBJECTS AND METHODS

Study type A prospective interventional randomized cohort study carried out at Critical Care Department, Cairo University Hospitals with 25 ICU beds for medical and surgical patients, in the period between December 2021 to January 2023.

An informed consent from 1st degree relatives was taken and confidentiality of information was assured.

Permission from the faculty of medicine ethical committee was obtained. Ethical committee approval number: MS-362-2019

Study design of the study population The patients' demographic data (including age, sex, baseline diseases, and causes of ICU admission) were extracted from their medical charts, and the patients' clinical characteristics (such as vital signs and hemodynamic parameters) were monitored as daily interval.

Laboratory data such as serum electrolyte concentrations, serum creatinine levels were extracted from the patients' medical charts.

Vit C level was measured for all patients (normal range 50-70 μM/L).

The patients' Acute Physiology and Chronic Health Evaluation II (APACHE II) and sequential organ failure assessment (SOFA) scores were calculated at the time of admission.

Patients were randomly divided into 2 groups into:

A) Treatment group (n=75) B) Control group (n=75) Ascorbic acid (Vitamin C) was given parenterally for the treatment group (2 gm every 8hrs) for 4 days.

Remeasuring the level of Vitamin C in all study population after 4 days.

• Measurement and administration of Vitamin C Vitamin C (Ascorbic Acid) parenteral formula Manufacturer: Arco Life sciences ( Http://www.arcolifesciences.co.in/ ) Ampules: each ampule contains 500 mg of ascorbic acid (5 ml each 1 ml contains 100mg) The dose and duration of intervention were selected based on the literature review.

Each dose of ascorbic acid was diluted in 50 ml of dextrose 5% solution and was administered as intravenous infusion over 30 minutes.

During the study period, patients were followed for any ascorbic acid-related adverse effects including nausea, vomiting, abdominal pain, hematuria, flushing, and significant arterial blood pressure change.

Measurement Kits This kit is an Enzyme-Linked Immunosorbent Assay (ELISA). The plate has been pre-coated with human Vitamin C antibody (VC). VC present in the sample is added and binds to antibodies coated on the wells. Substrate solution is then added and color develops in proportion to the amount of human VC and absorbance is measured at 450 nm.

* Manufacturer Bioassay Technology Labs
* Serial number: E1538Hu
* Standard Curve Range: 200 Mg/ml - 300 Mg/ml
* Sensitivity: 0.52 Mg/ml
* Size: 96 wells
* Storage: Store the reagents at 2-8°C. For over 6-month storage refer to the expiration date keep it at -20°C. Avoid repeated thaw cycles. If individual reagents are opened it is recommended that the kit be used within 1 month.
* Specimen Collection Serum Allow serum to clot for 10-20 minutes at room temperature. Centrifuge at 2000-3000 RPM for 20 minutes Plasma Collect plasma using EDTA or heparin as an anticoagulant. Centrifuge samples for 15 minutes at 2000-3000 RPM at 2 - 8°C within 30 minutes of collection.
* Calculation of results :

Plasma vitamin C level were measured by Vitamin C ELISA Kits by microgram /milliliter (μg/ml) and calculated to micromole/ L (μM/L) in factor of 5.6679 and results were given accordingly

• Normal range of Vitamin C in plasma : Multiple ranges are given in the level of vitamin C but recent studies consider range of (50-70μ M/L) is the reference in patients with sepsis and septic shock .

Statistical analysis Analysis of data was done using Statistical Program for Social Science version 20 (SPSS Inc., Chicago, IL, USA). Quantitative variables were described in the form of mean and standard deviation. Qualitative variables were described as number and percent. In order to compare parametric quantitative variables between two groups, Student t test was performed. Qualitative variables were compared using chi-square (X2) test or Fisher's exact test when frequencies were below five. Pearson correlation coefficients were used to assess the association between two normally distributed variables. When a variable was not normally distributed, A P value < 0.05 is considered significant The used tests were Chi-square test For categorical variables, to compare between different groups, Fisher's Exact or Monte Carlo correction for chi-square when more than 20% of the cells have expected count less than 5,Student t-test For normally distributed quantitative variables, to compare between two studied groups, ANOVA with repeated measures for normally distributed quantitative variables, to compare between more than two periods or stages, and Post Hoc test (Bonferroni adjusted) for pairwise comparisons, Pearson coefficient To correlate between two normally distributed quantitative variables, Mann Whitney test For abnormally distributed quantitative variables, to compare between two studied groups, Friedman test For abnormally distributed quantitative variables, to compare between more than two periods or stages and Post Hoc Test (Dunn's) for pairwise comparisons and Q: Cochran's test For non-parametric test for binary response variable and Post Hoc Test (Dunn's) for pairwise comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock (defined by sepsis induced hypotension i.e. MAP < 65 mmHg, tissue hypo-perfusion, vasopressors

Exclusion Criteria:

* Age below 18 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
C-reactive protein | Evaluated on a daily basis for 4 days
  C-reactive protein level III- Vasopressor (noradrenaline) dose and duration
Mean arterial blood pressure | Evaluated on a daily basis for 4 days
  Mean arterial blood pressure (MAP).

SECONDARY OUTCOMES:
ICU Length of stay . II- 7 day mortality rate. III- 28 days mortality | 28 days
  ICU Length of stay II- 7 day mortality rate. III- 28 days mortality
ICU mortality | 28 days
  ICU mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ashraf, MD, Study Director — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No